CLINICAL TRIAL: NCT07357636
Title: Longitudinal Cohort Study of Immune-Related Adverse Events in Solid Tumor Patients Receiving Immune Checkpoint Inhibitors, With Deep Phenotyping and Multi-Omics Biomarker Discovery
Brief Title: Longitudinal Cohort Study of Immune-Related Adverse Events in Solid Tumor Patients Treated With Immune Checkpoint Inhibitors
Status: Recruiting | Type: Observational
Sponsor: Shantou University Medical College (Other)
Collaborators: Fujian Medical University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Sun Yat-sen University (Other); Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Weidong Wang, Associate Professor, MD, Shantou University Medical College
Other Study IDs: 2023100
Record Dates: First submitted 2025-12-16; First posted 2026-01-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor; Immune-Related Adverse Events; Immunotherapy Toxicity
Keywords: Immune checkpoint inhibitors; Immunotherapy; Biomarkers; Neurotoxicity; Neuroimmune adverse events; immune related adverse events; PD-1 blocker
MeSH Terms: conditions — Neurotoxicity Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The study will retain a variety of biospecimens, including blood (whole blood, plasma, and serum), cerebrospinal fluid, urine, saliva, stool, gastric fluid, bile, synovial fluid, bronchoalveolar lavage fluid, pleural fluid, peritoneal lavage fluid, small intestinal fluid, colonic fluid, tears, tumor tissue, inflammatory biopsy tissue, matched normal tissue, pathology specimens (including formalin-fixed paraffin-embedded tissue), hair, and tongue coating samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Neuro-Sensory irAE Cohort: Participants who develop a grade ≥2 neurological, neurocognitive, psychiatric, ocular inflammatory, or peripheral nervous system immune-related adverse event.
- Gastrointestinal and Hepatic irAE Cohort: Participants who develop grade ≥2 immune-mediated colitis, hepatitis, pancreatitis, or related gastrointestinal toxicities.
- Rheumatology and Musculoskeletal irAE Cohort: Participants who develop grade ≥2 inflammatory arthritis, myositis, polymyalgia rheumatica-like syndromes, or related musculoskeletal toxicities.
- Vascular and Renal irAE Cohort: Participants who develop grade ≥2 myocarditis, vasculitis, nephritis, or other vascular or renal immune-mediated toxicities.
- Hematologic irAE Cohort: Participants who develop grade ≥2 immune-mediated cytopenias or other hematologic toxicities.
- Multi-Organ irAE Cohort: Participants who develop two or more distinct grade ≥2 immune-related adverse events involving different organ systems.
- Control Cohort: Participants who do not develop any grade ≥2 immune-related adverse events during the defined follow-up period.

SUMMARY:
Immune checkpoint inhibitors (ICIs) have transformed the treatment of solid tumors but are associated with immune-related adverse events (irAEs) that can affect virtually any organ system. While many irAEs are well recognized, neurological, neurocognitive, and psychiatric toxicities remain diagnostically challenging, potentially severe, and poorly understood, with limited predictive biomarkers.

This prospective longitudinal observational cohort study enrolls adult patients with solid tumors initiating a new course of ICI therapy. Participants undergo standardized baseline clinical assessments and biospecimen collection prior to ICI initiation, followed by longitudinal follow-up and event-driven sampling. Patients are dynamically assigned to organ-specific irAE cohorts based on the first clinically significant irAE that dictates management. Patients without grade ≥2 irAEs during follow-up serve as a comparator control cohort.

The primary objective is to characterize longitudinal immune and inflammatory biomarker trajectories associated with the development of irAEs and to identify predictive and prognostic biomarkers, with particular emphasis on neurological, neurocognitive, and psychiatric toxicities. Integrated clinical, imaging, and multi-omics data will be used to elucidate mechanisms of toxicity and inform future risk stratification and personalized management strategies.

DETAILED DESCRIPTION:
Immune checkpoint inhibitors targeting CTLA-4, PD-1, and PD-L1 pathways have demonstrated substantial clinical benefit across multiple solid malignancies. However, their mechanism of action can also lead to immune-related adverse events (irAEs), which may involve dermatologic, gastrointestinal, hepatic, pulmonary, endocrine, musculoskeletal, cardiovascular, renal, hematologic, neurological, and psychiatric systems. Neurological and neurocognitive irAEs, in particular, are uncommon but potentially devastating and remain poorly characterized.

This study is a hybrid prospective longitudinal observational cohort designed to move beyond reactive identification of irAEs toward proactive prediction and mechanistic understanding. Adult patients with solid tumors initiating a new ICI regimen are enrolled prior to treatment initiation. Longitudinal clinical data, imaging, and biospecimens are collected at predefined intervals and at the time of suspected irAE onset when feasible.

Participants are assigned to event-defined cohorts based on the first grade ≥2 irAE that drives clinical management, including neuro-sensory, gastrointestinal/hepatic, rheumatologic/musculoskeletal, vascular/renal, hematologic, multi-organ, or control (no significant irAE) cohorts. Deep phenotyping and multi-omics analyses-including immune cell profiling, proteomics, metabolomics, and microbiome analyses-are performed to identify biomarkers associated with irAE risk, severity, and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically confirmed solid malignancy
* Planned initiation of a new immune checkpoint inhibitor regimen (monotherapy or combination) as standard of care or on an approved clinical trial
* Ability to provide informed consent
* Baseline study assessments and biospecimen collection completed prior to first ICI dose
* Life expectancy of at least 6 months as determined by treating oncologist
* Availability of archival tumor tissue or willingness to undergo biopsy if archival tissue is unavailable

Exclusion Criteria:

* Uncontrolled medical, psychiatric, or social conditions that would interfere with study participation or data interpretation
* Chronic systemic immunosuppression exceeding 10 mg/day prednisone equivalent within 14 days prior to enrollment (excluding inhaled, topical, or physiologic replacement doses)
* Prior solid organ transplantation or allogeneic hematopoietic stem cell transplantation
* Untreated, symptomatic, or progressing brain metastases (treated and stable brain metastases allowed if off systemic steroids for at least 7 days)
* Inability or unwillingness to provide required baseline biospecimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) with histologically confirmed solid malignancies who are initiating a new immune checkpoint inhibitor regimen, either as standard of care or within an approved clinical trial. Participants are enrolled prior to the first immune checkpoint inhibitor dose and followed longitudinally to assess the development of immune-related adverse events and associated immune and inflammatory biomarker changes.
Sampling Method: Non-Probability Sample
Enrollment: 940 (Estimated)
Dates: Start 2019-01-10 (Actual); Primary Completion 2029-09-10 (Estimated); Study Completion 2029-09-10 (Estimated)

PRIMARY OUTCOMES:
Time to Clinical Resolution of Immune-Related Adverse Events (Days) | From irAE diagnosis through up to 24 months of follow-up
  Among participants who develop grade ≥2 immune-related adverse events (irAEs), the time from irAE diagnosis and initiation of organ-specific treatment (per institutional guidelines) to achievement of organ-specific clinical resolution will be recorded. Criteria for clinical resolution differ by organ system and are defined according to established consensus guidelines, as specified in the corresponding secondary outcome measures.

SECONDARY OUTCOMES:
Neuro-Sensory irAE Subgroup: Proportion of Participants with Modified Rankin Scale (mRS) Score ≤2 | 12 weeks after irAE diagnosis
  Among participants with immune-mediated neurological events (e.g., encephalitis, myelitis, plexopathy), functional status will be assessed using the Modified Rankin Scale. An mRS score ≤2 (slight disability, able to live independently) is a widely accepted threshold for favorable neurological outcome in neuroimmunology clinical trials.
Neuro-Sensory irAE Subgroup:Proportion of Participants with Objective Improvement on Nerve Conduction Studies | 12 weeks after irAE diagnosis
  Among participants with immune-mediated peripheral neuropathy, electrophysiologic improvement will be assessed using nerve conduction studies and electromyography. Objective improvement is defined as ≥20% improvement in motor or sensory nerve action potential amplitude or conduction velocity compared with the acute phase, according to EFNS/PNS criteria.
Psychiatric and Cognitive irAE Subgroup:Proportion of Participants with Patient Health Questionnaire-9 (PHQ-9) Score <10 | 8 weeks after initiation of targeted treatment
  Among participants with immune-mediated major depressive episodes, depressive symptoms will be assessed using the PHQ-9. A score <10 represents remission or mild symptoms and is an internationally accepted threshold distinguishing clinically significant depression from response/remission.
Psychiatric and Cognitive irAE Subgroup:Proportion of Participants with ≥0.5 Standard Deviation Improvement on ≥2 Standardized Neuropsychological Tests | 12 weeks after irAE diagnosis
  Among participants with immune-mediated cognitive impairment, standardized neuropsychological test batteries (including the Hopkins Verbal Learning Test-Revised and Trail Making Test Part B) will be administered. Clinically meaningful cognitive improvement is defined as ≥0.5 standard deviation improvement from the acute phase in at least two distinct cognitive domains.
Gastrointestinal and Hepatic irAE Subgroup: Proportion of Participants with ≤3 Bowel Movements per Day and No Hematochezia | 2 weeks after initiation of immunosuppressive therapy
  Among participants with immune-mediated colitis, clinical remission will be assessed. ≤3 bowel movements per day without hematochezia is a widely accepted clinical remission criterion in colitis clinical trials.
Gastrointestinal and Hepatic irAE Subgroup: Proportion of Participants with Alanine Aminotransferase (ALT) ≤1.5 × Upper Limit of Normal | 4 weeks after initiation of immunosuppressive therapy
  Among participants with immune-mediated hepatitis, biochemical remission will be assessed. ALT ≤1.5 × ULN is a commonly accepted biochemical remission criterion in drug-induced liver injury trials.
Rheumatologic and Musculoskeletal irAE Subgroup: Proportion of Participants with Clinical Disease Activity Index (CDAI) ≤10 | 12 weeks after initiation of immunosuppressive therapy
  Among participants with immune-mediated inflammatory arthritis, disease activity will be assessed using the CDAI. A CDAI score ≤10 defines low disease activity and is an established rheumatologic threshold.
Rheumatologic and Musculoskeletal irAE Subgroup: Proportion of Participants with ≥20% Improvement in Manual Muscle Testing (MMT-8) Score | 12 weeks after irAE diagnosis
  Among participants with immune-mediated myositis, muscle strength will be assessed using the MMT-8 score. A ≥20% improvement from the acute phase is an established clinically meaningful threshold in myositis trials.
Renal irAE Subgroup: Proportion of Participants with Serum Creatinine Recovery to Within 1.3 × Baseline | 12 weeks after irAE diagnosis
  Among participants with immune-mediated nephritis, renal recovery will be assessed. Serum creatinine recovery to within 1.3 × baseline represents a stringent and clinically meaningful recovery criterion per KDIGO acute kidney injury guidelines.
Hematologic irAE Subgroup: Proportion of Participants with Sustained Hematologic Response (CTCAE v5.0 Grade ≤1 for ≥4 Weeks) | Within 12 weeks after initiation of first-line immunosuppressive therapy
  Among participants with immune-mediated cytopenias, hematologic remission is defined as maintenance of CTCAE v5.0 grade ≤1 blood counts (e.g., platelets ≥75 ×10⁹/L, absolute neutrophil count ≥1.5 ×10⁹/L) for at least 4 weeks without ongoing transfusion or growth factor support.
Hematologic irAE Subgroup: Proportion of Participants with Normalized Lactate Dehydrogenase and Stable Hemoglobin | 2 weeks after initiation of treatment
  Among participants with immune-mediated hemolytic anemia, hemolysis control is defined as normalization of lactate dehydrogenase with stable hemoglobin levels for ≥7 days without transfusion support.
Multi-Organ irAE Subgroup: Proportion of Participants without Any New or Worsening ≥Grade 3 Immune-Related Adverse Events Across Organ Systems | Within 4 weeks after initiation of combined immunosuppressive therapy
  Among participants with multi-organ irAEs, overall toxicity control is defined as absence of any new or worsening grade ≥3 irAE in any organ system following initiation of treatment.
Multi-Organ irAE Subgroup: Proportion of Participants Requiring Intensive Care Unit Admission for Multi-Organ irAE | irAE diagnosis through resolution or up to 24 weeks
  The proportion of participants requiring intensive care unit admission due to the severity of multi-organ immune-related adverse events will be recorded as an objective marker of disease severity.
Control Cohort (No Grade ≥2 irAE): Duration of Immunotherapy without Grade ≥2 Immune-Related Adverse Events (Months) | From ICI initiation through 90 days after last dose
  Among participants who do not develop grade ≥2 irAEs, treatment tolerability will be assessed as the time from ICI initiation to first occurrence of grade ≥2 irAE, disease progression, death, or treatment discontinuation.
Control Cohort (No Grade ≥2 irAE): Proportion of Participants Completing Planned Immune Checkpoint Inhibitor Course per Protocol | From ICI initiation through 90 days after last dose
  Among participants without grade ≥2 irAEs, the proportion completing the planned ICI treatment course as scheduled will be recorded as a complementary measure of treatment tolerability.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Hainan Hospital of Chinese PLA General Hospital, Sanya
  - Affiliated Cancer Hospital of Shantou University Medical College, Shantou
  - the First Affiliated Hospital of Shantou University Medical College, Shantou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
1. Baseline Characteristics & Demographics: Age, sex, race/ethnicity, baseline body weight and height, diagnosis, treatment history, relevant comorbidities, smoking/alcohol status.
  2. Exposure/Treatment Data: Specific checkpoint inhibitor(s) received, dosing regimen, treatment start and end dates, medications.
  3. Laboratory & Diagnostic Data: Serial laboratory test results, key imaging findings relevant to irAEs, pathology reports.
  4. Outcomes: CTCAE grades, date to primary outcomes, management strategies.
  5. Oncologic Outcomes: Tumor response assessments.
  6. Supporting Documents for Data Interpretation.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2026.3 to 2029.1
Access Criteria: The de-identified IPD and supporting documents will be made available to qualified researchers worldwide upon request. Researchers will have access to the fully de-identified individual participant data listed in the previous section, along with the supporting documents including: the final study protocol, statistical analysis plan, the annotated case report forms. The data dictionary.
  All data will be anonymized in accordance with the HIPAA Safe Harbor method. Interested researchers must submit a formal research proposal outlining their study objectives, analysis plan, and ethical considerations via email for review by our Data Access Committee. Requestors will be required to sign a Data Use Agreement that legally binds them to use the data only for the approved purpose, maintain data security, and prevent re-identification or redistribution. Data will then be securely transferred via encrypted file sharing or made available through a controlled-access repository